CLINICAL TRIAL: NCT03533634
Title: Functional Outcome in Midshaft Clavicle Fracture Patients, Treated With Superior Versus Anteroinferior Reconstruction Plate. Randomized Clinical Trial.
Brief Title: Functional Outcome in Midshaft Clavicle Fracture, Treated With Superior Versus Anteroinferior Reconstruction Plate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMAE Hospital de Traumatologia y Ortopedia de Puebla (Other)
Responsible Party: Principal Investigator, Jose Antonio Manrique, Principal Investigator, UMAE Hospital de Traumatologia y Ortopedia de Puebla
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMAE
Record Dates: First submitted 2018-04-30; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Closed Fracture of Shaft of Clavicle
Keywords: midshaft clavicle fracture; functional outcome; anteroinferior plate; superior plate; reconstruction plate

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: the patient and the outcomes analyzer were masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- superior group (Experimental): this group with midshaft clavicle fracture were treated with superior reconstruction plate
  Interventions: Procedure: Open Reduction Internal Fixation superior plate
- anteroinferior group (Experimental): this group with midshaft clavicle fracture were treated with anteroinferior reconstruction plate
  Interventions: Procedure: Open Reduction Internal Fixation anteroinferior plate

INTERVENTIONS:
Procedure: Open Reduction Internal Fixation superior plate — 3.5mm superior reconstruction plate
  Arms: superior group
Procedure: Open Reduction Internal Fixation anteroinferior plate — 3.5mm anteroinferior reconstruction plate
  Arms: anteroinferior group

SUMMARY:
The purpose of this study was to evaluate the functional outcome in patients with a midshaft clavicle fracture treated with to different techniques. the first one was placing a 3.5mm reconstruction plate in the superior side of the clavicle and the second one placing the same 3.5mm reconstruction plate in the anteroinferior side of the clavicle. the patients had the same rehabilitation program and evaluated with functional scores at 30, 60, 90 and 365 days after surgery. biomechanical studies have demonstrated more stable construct using an anteroinferior plate in clavicle fractures and we were trying to find out if it has a clinical relevance in patients with midshaft clavicle fractures.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the functional outcome in patients with a midshaft clavicle fracture treated with to different techniques.

the first technique was placing a 3.5mm reconstruction plate in the superior side of the clavicle and the second one placing the same 3.5mm reconstruction plate in the anteroinferior side of the clavicle.

the patients had the same rehabilitation program and evaluated with Disabilities Arm Shoulder and Hand functional outcome score and Visual Analogue Score for pain at 30, 60, 90 and 365 days after surgery.

biomechanical studies have demonstrated more stable construct using an anteroinferior plate in clavicle fractures and we were trying to find out if it has a clinical relevance in patients with midshaft clavicle fractures.

ELIGIBILITY:
Inclusion Criteria:

* traumatic fracture
* ao 15 b1 and 15 b2
* no previous shoulder lesions
* no further 7 days fractures
* closed fracture

Exclusion Criteria:

* calcium diseases
* Previous shoulder pain
* other fractures associated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Disabilities of Arm Shoulder and Hand score (DASH) | 30 days after surgery
  we applied the Disabilities of arm, shoulder and hand score a score from 0 to 100 where 0 is no disability and 100 the worst disability
Disabilities of Arm Shoulder and Hand score (DASH) | 60 days after surgery
  we applied the Disabilities of arm, shoulder and hand score a score from 0 to 100 where 0 is no disability and 100 the worst disability
Disabilities of Arm Shoulder and Hand score (DASH) | 90 days after surgery
  we applied the Disabilities of arm, shoulder and hand score a score from 0 to 100 where 0 is no disability and 100 the worst disability
Disabilities of Arm Shoulder and Hand score (DASH) | 365 days after surgery
  we applied the Disabilities of arm, shoulder and hand score a score from 0 to 100 where 0 is no disability and 100 the worst disability

SECONDARY OUTCOMES:
Visual Analogue Scale score (VAS) | 30 days after surgery
  we applied Visual Analogous Scale pain score a 0 to 10 score where 0 is no pain and 10 the maximum grade of pain
Visual Analogue Scale score (VAS) | 60 days after surgery
  we applied Visual Analogous Scale pain score a 0 to 10 score where 0 is no pain and 10 the maximum grade of pain
Visual Analogue Scale score (VAS) | 90 days after surgery
  we applied Visual Analogous Scale pain score a 0 to 10 score where 0 is no pain and 10 the maximum grade of pain
Visual Analogue Scale score (VAS) | 365 days after surgery
  we applied Visual Analogous Scale pain score a 0 to 10 score where 0 is no pain and 10 the maximum grade of pain

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Manrique, MD, Principal Investigator — UMAE Hospital de Traumatologia y Ortopedia de Puebla; Gustavo Rivera Saldivar, MD, Study Chair — UMAE Hospital de Traumatologia y Ortopedia de Puebla

IPD SHARING:
Plan to Share IPD: Undecided